CLINICAL TRIAL: NCT05009979
Title: 18F-DCFPyL PET/CT in Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reason for termination was a combination of slow accrual in setting of austerity measures regarding resource allocation.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Esther Mena, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000080; 000080-C
Record Dates: First submitted 2021-08-17; First posted 2021-08-18 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Imaging; Liver Cancer; Radiotracer; PSMA
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Imaging; Tomography, X-Ray Computed; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1, Cohort 1 Baseline and Post-treatment Imaging with Piflufolastat F-18 (18F-DCFPyL) (Experimental): Piflufolastat F-18 (18F-DCFPyL) positron emission tomography computed tomography (PET/CT) imaging, CT and/or magnetic resonance imaging (MRI) and standard of care local ablative treatment
  Interventions: Drug: F18-FDG; Device: MRI; Device: CT; Drug: F18-DCFPyL; Procedure: Tumor biopsy

INTERVENTIONS:
Drug: F18-FDG — Within approximately 2 weeks of each piflufolastat F-18 (18F-DCFPyL) positron emission tomography/ computed tomography (PET/CT) scan, participants will be scanned with a fludeoxyglucose F 18 (18F-FDG) PET/CT imaging at the NIH Clinical Center using standard procedures. The 18F-FDG PET/CT imaging performed will allow the localization of viable tumor sites and characterize their FDG metabolism for comparison with 18F-DCFPyL imaging. The 18F-FDG PET/CT imaging will consist of an 18F-FDG injection and PET/CT imaging performed approximately 1 hour post 18F-FDG injection. A corresponding low dose CT scan for attenuation correction and co-registration purposes will be performed prior to the PET image.
  Other Names: Fludeoxyglucose F 18
Device: MRI — A standard of care computed tomography (CT) and/or magnetic resonance imaging (MRI) will be performed within 2 months of each piflufolastat F-18 (18F-DCFPyL) positron emission tomography (PET/CT).
  Other Names: Magnetic resonance imaging
Device: CT — A standard of care computed tomography (CT) and/or magnetic resonance imaging (MRI) will be performed within 2 months of each piflufolastat F-18 (18F-DCFPyL) positron emission tomography (PET/CT).
  Other Names: Computed tomography
Drug: F18-DCFPyL — Each subject will receive a single intravenous (IV) dose of piflufolastat F-18 (18F-DCFPyL) by bolus injection at a rate of approximately 1 ml/3-5 sec. The maximum amount of injected active drug will be less than 4.02 microgram. The target administered activity will be 9 mCi. The 18F-DCFPyL positron emission tomography and computed tomography (PET/CT) imaging will consist of the 18F-DCFPyL injection, followed by approximately 45 min dynamic CT imaging of a single bed position (including the liver lesion), and a static whole-body PET/CT imaging (top of head to mid-thighs) performed at 1 hour (+/-10 minutes) post 18F-DCFPyL injection. Only a single injection of 18F-DCFPyL is required. The initial 45 minutes dynamic regional scan will be used to determine the kinetics of 18F-DCFPyL within the tumor as compared with normal liver and other background.
  Other Names: piflufolastat F-18
Procedure: Tumor biopsy — Principal investigator discretion pre-treatment or during surgical resection.

SUMMARY:
Background:

A radiotracer (or tracer) is a radioactive substance. It is used in Positron Emission Tomography (PET) imaging to help see specific sites in the body. Researchers want to learn if a new tracer can help them better identify hepatocellular cancer (HCC) in people.

Objective:

To learn if a radiotracer called piflufolastat F-18 (18F-DCFPyL), can identify sites of HCC better than current standard imaging.

Eligibility:

Adults aged 18 years and older who may have HCC based on previous standard imaging.

Design:

Participants will be screened with a medical history, physical exam, and blood tests. They will have a computed tomography (CT) and/or magnetic resonance imaging (MRI) scan.

Participants will have a whole-body positron emission tomography (PET/CT) scan. The PET and CT scanners use x-rays to make pictures of the inside of the body. The PET uses a tracer to help make the pictures. Participants will get an intravenous (IV) injection of 18F-DCFPyL 1 hour before the scan.

Within two weeks, participants will have a Fludeoxyglucose F 18 (18F-FDG) PET/CT scan. 18F-FDG is a commonly used tracer. They will get 18F-FDG via IV 1 hour before the scan.

Participants will have a CT/magnetic resonance imaging (MRI) within 2 months of the first 18F-DCFPyL PET/CT.

Participants will have standard treatment for their cancer. During treatment, they will have a tumor biopsy. If the biopsy shows they do not have HCC, they will be removed from the study.

For participants who have HCC and their cancer was identified in the 18F-DCFPyL PET/CT, they will have a second 18F-DCFPyL PET/CT and 18F-FDG PET/CT.

Participants will have follow-up visits every 3 months for 2 years. Then they will have yearly visits for 3 years.

DETAILED DESCRIPTION:
Background:

Prostate specific membrane antigen is overexpressed in high-grade tumors, and increases when de-differentiation, metastatic or hormone-refractory disease occur, making the expression level a prognostic factor for disease outcome.

It has been shown that prostate-specific membrane antigen (PSMA) can be expressed not only on prostate cancer cells, but also on cell lines of other malignancies, as well as tumor endothelium.

A recent publication reported that nearly 95% of hepatocellular carcinoma (HCC) stained positive for PSMA in the tumor vasculature. Research suggests that the process of endothelial cell recruitment to HCC occurs early and throughout the process of hepatic tumorigenesis, making an endothelial cell tracer an ideal marker to detect early disease.

18F-DCFPyL, a second generation PSMA PET agent, binds with high affinity to PSMA yet clears rapidly from the blood pool and thus, whole-body PET imaging with this agent, may provide a new tool in staging high risk cancers and detecting recurrent disease.

We propose to expand our clinical work using 18F-DCFPyL and evaluate its usefulness for detecting sites of hepatocellular carcinoma.

Objective:

To assess the ability of 18F-DCFPyL PET/CT imaging to detect sites of hepatocellular carcinoma

Eligibility:

Participants >= 18 years old

High radiological suspicion of hepatocellular carcinoma (HCC) with at least one measurable lesion on standard imaging modality (CT and/or MRI)

Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2

Design:

This is a multi-site imaging study enrolling participants with suspected hepatocellular carcinoma. The accrual ceiling is set to 50 participants.

All participants will undergo a baseline 18F-DCFPyL PET/CT scan. A standard of care CT and/or MRI will be performed within 2 months of the 18F-DCFPyL PET/CT. Participants will be also scanned with an 18F-FDG PET/CT imaging within approximately 2 weeks of the 18F-DCFPyL PET/CT imaging.

Participants will be scheduled to undergo a biopsy prior to or during standard of care local treatment for HCC (e.g., resection, radiofrequency ablation, microwave ablation, transarterial embolization (TAE), stereotactic body radiotherapy (SBRT)).

Participants with a baseline positive 18F-DCFPyL-PET/CT imaging (i.e. with the presence of DCFPyL-avid tumor/s) and biopsy confirming HCC diagnosis will undergo a post-treatment 18F-DCFPyL PET/CT imaging during the first routine follow-up period, typically within 16 weeks. Subjects with negative tumor uptake at baseline 18F-DCFPyL-PET/CT will not be re-scanned post-treatment but will remain in follow-up.

Participants with a positive HCC biopsy will be followed for 5 years to assess progression free survival.

ELIGIBILITY:
* INCLUSION CRITERIA:
* High radiological suspicion of hepatocellular carcinoma (LR4 (probably hepatocellular carcinoma) or LR5 (definitely hepatocellular carcinoma) based on the most current version of Liver Imaging Reporting & Data System (LI-RADS) with at least one measurable lesion on standard imaging modality computed tomography (CT) and/or magnetic resonance imaging (MRI).
* Eligible for local therapies (included but not limited to surgical resection, stereotactic radiation therapy, transarterial chem/radio/bland embolization, microwave ablation, radiofrequency ablation).
* Ability to take oral medication and be willing to adhere to the study intervention regimen.
* Age >=18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.
* Known human immunodeficiency virus (HIV)-infected individuals must be on effective anti-retroviral therapy with undetectable viral load within 6 months.
* Known chronic hepatitis B virus (HBV) infected individuals, must be on suppressive therapy with undetectable viral load.
* Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured.
* The effects of piflufolastat F-18 (18F-DCFPyL) (study drug) on the developing human fetus are unknown. For this reason and because this agent as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 2 months after each study positron emission tomography and computed tomography (PET/CT) imaging. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-DCFPyL, or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics.
* Other medical conditions deemed by the principal investigator (or associates) to make the subject unsafe/ineligible for protocol procedures.
* Subjects weighing > 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry
* Serum creatinine > 2 times the upper limit of normal
* Pregnant women are excluded from this study because 18F-DCFPyL is an agent with the potential for teratogenic or abortifacient effects. as well as other agents used in this trial are known to be teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Mena Gonzalez, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data is available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data is made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Mena E, Shih J, Chung JY, Jones J, Rabiee A, Monge C, Turkbey B, Lindenberg L, Salerno KE, Kassin M, Wood B, Hernandez J, Maass-Moreno R, Saboury B, Jakhete N, Molitoris JK, Unger KR, Choyke PL, Escorcia FE. Functional Imaging of Liver Cancer (FLIC): Study protocol of a phase 2 trial of 18F-DCFPyL PET/CT imaging for patients with hepatocellular carcinoma. PLoS One. 2022 Nov 11;17(11):e0277407. doi: 10.1371/journal.pone.0277407. eCollection 2022. PMID 36367894
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000080-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1, Cohort 1 Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL): Participants with radiographically confirmed hepatocellular carcinoma. Piflufolastat F-18 (18F-DCFPyL) positron emission tomography and computed tomography (PET/CT) imaging, CT and/or magnetic resonance imaging (MRI) and standard of care local ablative treatment F18-FDG: Within approximately 2 weeks of each piflufolastat F-18 (18F-DCFPyL) positron emission tomography and computed tomography (PET/CT) scan, participants will be scanned with a fludeoxyglucose F 18 (18F-FDG) PET/CT imaging at the National Institutes of Health (NIH) Clinical Center using standard procedures. The 18F-FDG PET/CT imaging performed will allow the localization of viable tumor sites and characterize their fludeoxyglucose-18 (FDG) metabolism for comparison with 18F-DCFPyL imaging. The 18F-FDG PET/CT imaging will consist of an 18F-FDG injection and PET/CT imaging performed approximately 1 hour post 18F-FDG injection. A corresponding low dose CT scan for attenuation correction and co-registration purposes will be performed prior to the PET image.
Period: Overall Study
Arm/Group | Arm 1, Cohort 1 Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL): Participants with radiographically confirmed hepatocellular carcinoma. Piflufolastat F-18 (18F-DCFPyL) positron emission tomography and computed tomography (PET/CT) imaging, CT and/or magnetic resonance imaging (MRI) and standard of care local ablative treatment F18-FDG: Within approximately 2 weeks of each piflufolastat F-18 (18F-DCFPyL) positron emission tomography and computed tomography (PET/CT) scan, participants will be scanned with a fludeoxyglucose F 18 (18F-FDG) PET/CT imaging at the National Institutes of Health (NIH) Clinical Center using standard procedures. The 18F-FDG PET/CT imaging performed will allow the localization of viable tumor sites and characterize their fludeoxyglucose-18 (FDG) metabolism for comparison with 18F-DCFPyL imaging. The 18F-FDG PET/CT imaging will consist of an 18F-FDG injection and PET/CT imaging performed approximately 1 hour post 18F-FDG injection. A corresponding low dose CT scan for attenuation correction and co-registration purposes will be performed prior to the PET image.
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.75 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) Defined as the Proportion of Histopathology Positive Lesions as Measured by the Maximum Standardized Uptake (SUVmax) Value
Description: Positive predictive value is defined as the proportion of histopathologically positive lesions. Positron emission tomography (PET) positivity was measured by the maximum standardized uptake (SUVmax) value. The 95% confidence intervals of the positive predictive value of piflufolastat F-18 (18F-DCFPyL) positron emission tomography scan and computed tomography (PET/CT) will be reported in which the confidence limits are the 2.5th and 97.5th percentile of the 2000 bootstrap samples obtained by random sample without replacement at the participant level to account for inter-lesion correlation. For lesions within the liver, a focal abnormal area of increased 18F-DCFPyL activity higher than the surrounding liver uptake (SUVmax more than x 1.2 times than the normal liver-SUV mean) will be considered positive. For lesions outside the liver, a positive lesion is defined as focal abnormal uptake higher than the blood pool or surrounding normal organ or soft tissue background.
Time Frame: Baseline, post ablation, and disease progression, an average of 3.87 months
Population: 7/8 participants were analyzed because one participant only completed baseline fludeoxyglucose-18 (FDG) PET/CT but did not undergo baseline 18F-DCFPyL or post treatment PET/CT scans. No biopsies at post ablation, and outside the liver were collected because this intervention was not part of the study. No participants had disease progression while on study, therefore no biopsies were collected. We did not scan participants with 18F-DCFPyL at progression/no signs of progression while on study.
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: lesions
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
Number analyzed (lesions) | 8
proportion of lesions
  Lesions within the liver at baseline | 0.875 [0.64 to 1.10]
  Lesions within the liver post ablation: number analyzed (Participants) | 0
  Lesions within the liver post ablation: number analyzed (lesions) | 0
  Lesions within the liver at disease progression: number analyzed (Participants) | 0
  Lesions within the liver at disease progression: number analyzed (lesions) | 0
  Lesions outside the liver at baseline: number analyzed (Participants) | 0
  Lesions outside the liver at baseline: number analyzed (lesions) | 0
  Lesions outside the liver post ablation: number analyzed (Participants) | 0
  Lesions outside the liver post ablation: number analyzed (lesions) | 0
  Lesions outside the liver at disease progression: number analyzed (Participants) | 0
  Lesions outside the liver at disease progression: number analyzed (lesions) | 0

2. Primary Outcome: Point Estimates of the Positive Predictive Value of Piflufolastat F-18 (18F-DCFPyL)
Description: Positive predictive value of the DCFPyL PET imaging agent is defined as the proportion of radiologically positive lesions (true positives) that were PET positive, over the radiologically (CT/MRI) positive lesions that were PET positive (true positives) added to the radiologically negative lesions that were PET positive (false positives). Point estimates and 95% confidence intervals of the positive predictive values of piflufolastat F-18 (18F-DCFPyL) positron emission tomography scan and computed tomography (PET/CT) will be reported in which the confidence limits are the 2.5th and 97.5th percentile of the 2000 bootstrap samples obtained by random sample without replacement at the participant level to account for inter-lesion correlation.
Time Frame: Baseline, post ablation, disease progression, an average of 3.87 months
Population: 7/8 participants were analyzed because one participant only completed baseline fludeoxyglucose-18 (FDG) PET/CT but did not undergo baseline 18F-DCFPyL or post treatment PET/CT scans. No biopsies at post ablation were collected because this intervention was not part of the study. No participants had disease progression while on study, therefore no biopsies were collected.
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: lesions
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
Number analyzed (lesions) | 14
proportion of lesions
  Baseline | 0.64 [0.39 to 0.89]
  Post ablation: number analyzed (Participants) | 0
  Post ablation: number analyzed (lesions) | 0
  Disease progression: number analyzed (Participants) | 0
  Disease progression: number analyzed (lesions) | 0

3. Secondary Outcome: Lesion Level Sensitivity
Description: Lesion level sensitivity is defined as true positive (TP)/[TP+ false negative (FN], being TP = true positive lesions (i.e., positron emission tomography (PET) positive lesions that are histologically positive) and FN = false negative lesions (i.e., PET negative lesions that are histologically positive) . The lesion level sensitivity of piflufolastat F-18 (18F-DCFPyL) positron emission tomography scan and a computed tomography (PET/CT) and CT/magnetic resonance imaging (MRI) will be calculated and compared. The confidence interval for each estimate will be obtained from the bootstrap samples and the difference in the estimates between the imaging modalities will be compared by the Wald test with the standard error calculated from the bootstrap samples.
Time Frame: Baseline, post ablation, and disease progression, an average of 3.87 months
Population: 7/8 participants were analyzed because one participant only completed baseline fludeoxyglucose-18 (FDG) PET/CT but did not undergo baseline 18F or post treatment PET/CT scans. No biopsies at post ablation were collected because this intervention was not part of the study or standard of care. No data is available at disease progression because none of the participants showed signs of disease progression while on study.
Measure: Number (95% Confidence Interval); unit: proportion of biopsy lesions
Units Other Than Participants: lesions
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
Number analyzed (lesions) | 14
proportion of biopsy lesions
  Sensitivity with CT/MRI at baseline | 1.0 [1.0 to 1.0]
  Sensitivity with CT/MRI at CT/MRI post ablation: number analyzed (Participants) | 0
  Sensitivity with CT/MRI at CT/MRI post ablation: number analyzed (lesions) | 0
  Sensitivity with CT/MRI at disease progression: number analyzed (Participants) | 0
  Sensitivity with CT/MRI at disease progression: number analyzed (lesions) | 0
  Sensitivity with 18F-DCFPyL PET/CT at baseline | 0.87 [0.70 to 1.04]
  Sensitivity with 18F-DCFPyL PET/CT post ablation: number analyzed (Participants) | 0
  Sensitivity with 18F-DCFPyL PET/CT post ablation: number analyzed (lesions) | 0
  Sensitivity with 18F-DCFPyL PET/CT at disease progression: number analyzed (Participants) | 0
  Sensitivity with 18F-DCFPyL PET/CT at disease progression: number analyzed (lesions) | 0

4. Secondary Outcome: Lesion Level Specificity
Description: Lesion level specificity is defined as true negative (TN)/[TN+ false positive (FP], being TN = true negative (i.e., positron emission tomography (PET) negative lesions that are histopathologically negative, and FP = false positive (i.e., PET positive lesions that are histopathologically negative). The lesion level specificity of piflufolastat F-18 (18F-DCFPyL) positron emission tomography scan and a computed tomography (PET/CT) and CT/magnetic resonance imaging (MRI) will be calculated and compared. The confidence interval for each estimate will be obtained from the bootstrap samples and the difference in the estimates between the imaging modalities will be compared by the Wald test with the standard error calculated from the bootstrap samples.
Time Frame: Baseline, post ablation, and disease progression, an average of 3.87 months
Population: No biopsies at post ablation were collected because this intervention was not part of the study or standard of care. No data is available at disease progression because none of the participants showed signs of disease progression while on study.
Measure: Number (95% Confidence Interval); unit: proportion of biopsy lesions
Units Other Than Participants: lesions
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
Number analyzed (lesions) | 14
proportion of biopsy lesions
  Specificity with CT/MRI at baseline | NA [NA to NA] — Specificity can't be calculated because there are no true negative lesions since biopsies were not performed in non-malignant lesions.
  Specificity with CT/MRI post ablation: number analyzed (Participants) | 0
  Specificity with CT/MRI post ablation: number analyzed (lesions) | 0
  Specificity with CT/MRI at disease progression: number analyzed (Participants) | 0
  Specificity with CT/MRI at disease progression: number analyzed (lesions) | 0
  Specificity with 18F-DCFPyL PET/CT at baseline | NA [NA to NA] — Specificity can't be calculated because there are no true negative lesions since biopsies were not performed in non-malignant lesions.
  Specificity with 18F-DCFPyL PET/CT post ablation: number analyzed (Participants) | 0
  Specificity with 18F-DCFPyL PET/CT post ablation: number analyzed (lesions) | 0
  Specificity with 18F-DCFPyL PET/CT at disease progression: number analyzed (Participants) | 0
  Specificity with 18F-DCFPyL PET/CT at disease progression: number analyzed (lesions) | 0

5. Secondary Outcome: Lesion Level Positive Predictive Value
Description: Lesion level positive predictive value is defined as true positive (TP/[TP+ false positive (FP], being TP = true positive (i.e., positron emission tomography (PET) positive lesions that are histopathologically positive) and FP = false positive (i.e., PET positive lesions that are histopathologically negative) . The lesion level positive predictive value of piflufolastat F-18 (18F-DCFPyL) positron emission tomography scan and a computed tomography (PET/CT) and CT/magnetic resonance imaging (MRI) will be calculated and compared. The confidence interval for each estimate will be obtained from the bootstrap samples and the difference in the estimates between the imaging modalities will be compared by the Wald test with the standard error calculated from the bootstrap samples.
Time Frame: Baseline, post ablation, and disease progression, an average of 3.87 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of biopsy lesions
Units Other Than Participants: lesions
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
Number analyzed (lesions) | 14
proportion of biopsy lesions
  Positive Predictive Value with CT/MRI at baseline | 0.57 [0.31 to 0.83]
  Positive Predictive Value with CT/MRI post ablation: number analyzed (Participants) | 0
  Positive Predictive Value with CT/MRI post ablation: number analyzed (lesions) | 0
  Positive Predictive Value with CT/MRI at disease progression: number analyzed (Participants) | 0
  Positive Predictive Value with CT/MRI at disease progression: number analyzed (lesions) | 0
  Positive Predictive Value with 18F-DCFPyL PET/CT at baseline | 0.50 [0.23 to 0.76]
  Positive Predictive Value with 18F-DCFPyL PET/CT post ablation: number analyzed (Participants) | 0
  Positive Predictive Value with 18F-DCFPyL PET/CT post ablation: number analyzed (lesions) | 0
  Positive Predictive Value with 18F-DCFPyL PET/CT at disease progression: number analyzed (Participants) | 0
  Positive Predictive Value with 18F-DCFPyL PET/CT at disease progression: number analyzed (lesions) | 0

6. Secondary Outcome: Change in Piflufolastat F-18 (18F-DCFPyL) Positron Emission Tomography and Computed Tomography (PET/CT) Maximum Standardized Uptake Value (SUVmax) Between Pre- and Post-treatment
Description: Change in 18F-DCFPyL PET/CT maximum standardized uptake value (SUVmax) between pre- and post-treatment tumor or tumor bed will be compared by paired Wilcoxon test for participants who undergo local treatment for hepatocellular carcinoma. Positive uptake is defined as a focal abnormal area of increased 18F-DCFPyL activity higher than the surrounding liver uptake standard update value (SUV)max more than x 1.2 times than the normal liver-SUV mean). Negative uptake is defined as tumor uptake less than adjacent background soft tissue, or less than blood pool for lymph nodes.
Time Frame: Pre- and post-treatment hepatocellular carcinoma (HCC) 18F-DCFPyL PET scans, an average of 3.2 months.
Population: 7/8 participants were analyzed because one participant only completed baseline fludeoxyglucose-18 (FDG) PET/CT but did not undergo baseline 18F-DCFPyL or post treatment PET/CT scans.
Measure: Mean (95% Confidence Interval); unit: SUV
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 7
SUV
  Tumor pre-treatment | 10.72 [1.88 to 12.60]
  Tumor post-treatment | 4.61 [2.34 to 6.87]
  Tumor bed pre-treatment | 10.72 [1.88 to 12.60]
  Tumor bed post-treatment | 4.61 [2.34 to 6.87]

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Document adverse events from the first study intervention through 3 days after the agent was last administered, an average of 3.87 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
Number analyzed (Participants) | 8
Participants | 7

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 3.87 months. Adverse Events were monitored/assessed from the first study intervention through 3 days after the agent was last administered, an average of 3.87 months.
Arm/Group | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL) (N=8)
Ascites (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Baseline and Post-treatment Imaging With Piflufolastat F-18 (18F-DCFPyL) (N=8)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
White blood cell decreased (Investigations) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol 000080-C version date 120123 (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05009979/Prot_SAP_000.pdf
  • Study Protocol: Protocol 000080-C NIH Addendum version date 120123 (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05009979/Prot_001.pdf
  • Informed Consent Form (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT05009979/ICF_002.pdf